CLINICAL TRIAL: NCT01670357
Title: Placebo Controlled, Dose-Response, Randomized, Double Blind, Phase II Study to Evaluate the Efficacy and Safety of DA-6034 Eye Drops in Patients With Dry Eye Syndrome
Brief Title: Phase II Study of DA-6034 Eye Drops in Dry Eye Syndrome
Acronym: DES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DA6034_DES_II
Record Dates: First submitted 2012-01-19; First posted 2012-08-22 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes | interventions — recoflavone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- DA-6034 Low dose (Experimental): DA-6034 3%
  Interventions: Drug: DA-6034 3%
- DA-6034 High dose (Experimental): DA-6034 5%
  Interventions: Drug: DA-6034 5%
- Placebo (Placebo Comparator): DA-6034 Placebo
  Interventions: Drug: DA-6034 Placebo

INTERVENTIONS:
Drug: DA-6034 3% — Eye drop, 1 drop/each eye, 4 times/day, for 4 weeks
  Other Names: DA-6034 Low dose
  Arms: DA-6034 Low dose
Drug: DA-6034 5% — Eye drop, 1 drop/each eye, 4 times/day, for 4 weeks
  Other Names: DA-6034 High dose
  Arms: DA-6034 High dose
Drug: DA-6034 Placebo — Eye drop, 1 drop/each eye, 4 times/day, for 4 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This study is to determine the efficacy and safety of 3% or 5% DA-6034 eye drops compared with placebo in dry eye syndrome.

DETAILED DESCRIPTION:
Eligible subjects are randomly assigned to receive 3% DA-6034, 5% DA-6034 or Placebo. This study is conducted for 6 weeks(Run-in Period 2 weeks + Treatment Period 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Age≥20
2. Dry eye symptoms(irritation, foreign body sensation, burning, mucus discharge, blurring, itching, photophobia, tird or heavy feeling, pain) for more than 6 months
3. Fluorescein corneal staining score ≥ 4 and Schirmer test I ≤ 7mm in same eye
4. Corrected vision ≥ 0.2 in both eye
5. Have given a written, informed consent

Exclusion Criteria:

1. Ocular disorder that may confound interpretation of study results
2. Current treatment for glaucoma or IOP over 25mmHg
3. Ocular surgery history within 1 year
4. Other malignancy history or uncontrolled severe disease within 5 years
5. Use of systemic immunosuppressive therapies within 3 months
6. Use of opthalmic cyclosporin, opthalmic steroid within 4 weeks
7. Received any other investigational drugs within 4 weeks
8. Subjects who are willing to wear contact lenses during study participation
9. Pregnant or lactating women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Fluorescein Corneal Staining(FCS) score | 4 weeks
  Change from baseline means the change between 0 weeks and 4 weeks.

SECONDARY OUTCOMES:
Change from baseline of Tear Break-Up Time(TBUT) | 4 weeks
  Change from baseline means the change between 0 weeks and 4 weeks.
Change from baseline of Lissamine Green Conjunctival Staining(LGCS) score | 4 weeks
  Change from baseline means the change between 0 weeks and 4 weeks.
Change from baseline of Schirmer Test I score | 4 weeks
  Change from baseline means the change between 0 weeks and 4 weeks.
Change from baseline of Ocular Surface Disease Index(OSDI) score | 4 weeks
  Change from baseline means the change between 0 weeks and 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: ManSoo Kim, M.D., Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St.Mary's hospital, Seoul, South Korea